CLINICAL TRIAL: NCT04909073
Title: An Observational Study of Afatinib 30 mg Daily in Patients With Advanced Non-small Cell Lung Cancer (NSCLC) Harbouring Common EGFR Mutations Treated With Afatinib
Brief Title: Observational Study of Afatinib 30 mg Daily
Status: Recruiting | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.0303
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer; Epidermal Growth Factor Receptor Mutation
Keywords: afatinib; EGFR mutation-positive NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Afatinib 30 mg daily: Oral afatinib 30 mg tablet once daily, continuously
  Interventions: Drug: Afatinib

INTERVENTIONS:
Drug: Afatinib — Continuous treatment of afatinib 30mg tablet once daily in the absence of disease progression or unacceptable treatment-related toxicity, Investigator decision or patient decision to discontinue study treatment.
  Other Names: Giotrif

SUMMARY:
Afatinib, a first-in-class irreversible ErbB family blocker, is a 1st line treatment option for patients with advanced stage NSCLC harbouring sensitizing EGFR mutations. In randomized 1st line studies of afatinib at a standard dose of 40 mg daily versus standard of care, 28-53% of patients required a dose reduction due to adverse events (AE) induced by afatinib. The most common AEs are cutaneous and gastrointestinal (diarrhoea, dysphagia, and mucositis). Prevalence of diarrhoea in patients receiving 40 mg of afatinib, in 1st line phase II and III studies is as high as 90.0% (all grades of diarrhoea) and 14.4% (grade 3-4 diarrhoea). Another important gastrointestinal AE is mucositis, which presents in 51.9%-64.4% of patients treated with afatinib, with only 4.4%-8.3% of the cases being grade 3-4. Dose reduction tended to occur in patients who had higher initial afatinib plasma concentrations and led to decreases in the incidence and severity of afatinib-related AEs without affecting therapeutic efficacy. The incidence of gastrointestinal AEs could be decreased >50% with proper afatinib dose reduction.

The effect of 1st line afatinib 30 mg daily in patients with EGFR mutation-positive NSCLC is unknown. We hypothesize that, in patients with EGFR mutation-positive NSCLC, 1st line afatinib treatment at 30 mg daily is tolerable with less gastrointestinal AEs and with a similar efficacy to standard dose afatinib.

DETAILED DESCRIPTION:
This is a multi-country, multi-centre, study designed to collect clinical data and to evaluate efficacy and safety of patients treated with afatinib 30 mg at the Investigator's discretion.

All entered patients (i.e., patients that have been treated with the defined medication) will receive continuous treatment of afatinib in the absence of disease progression or meeting any other withdrawal criteria. All patients will visit Investigator at regular intervals for assessment of efficacy and safety as outlined in the Flow Chart for the first 7 cycles treatment. The Investigator will assess the patient at each visit. Tumour response and progression will be assessed using RECIST 1.1 at the Investigator site.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. ECOG performance status 0-1.
3. Pathologically confirmed diagnosis of Stage IIIB/IV adenocarcinoma of the lung.
4. Have been commenced on first line afatinib 30 mg within 4 weeks of study enrolment.
5. Documented EGFR mutation(s)-positive NSCLC (common mutations: Del19 and L858R) from tumour biopsy material. Results of EGFR mutation test must be available before taking Afatinib.
6. A CT thorax/ abdomen within 4 weeks of study enrolment with at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumours (RECIST) version 1.1.
7. No brain metastases (confirmed by a CT or MRI brain performed within 4 weeks of study enrolment)
8. Documented adequate organ function before taking Afatinib:

   * Absolute neutrophil count (ANC) ≥1500/mm3. (ANC >1000/mm3 may be considered in special circumstances such as benign cyclical neutropenia as judged by the Investigator and in discussion with the sponsor-Investigator).
   * Platelet count ≥75,000/mm3.
   * Estimated creatinine clearance using Cockcroft Gault calculation of at least 45 ml/min.
   * Total Bilirubin ≤1.5 times upper limit of (institutional/central) normal (Patients with Gilbert's syndrome total bilirubin must be ≤4 times institutional upper limit of normal).
   * Aspartate amino transferase (AST) or alanine amino transferase (ALT) ≤3 times the upper limit of (institutional/central) normal (ULN) (if related to liver metastases ≤5 times ULN).
9. Archived tissue sample is available.
10. Written informed consent per regulations.

Exclusion Criteria:

1. Prior chemotherapy for Stage IIIB/IV adenocarcinoma of the lung. Neo-/adjuvant chemotherapy, CT-RT or RT is permitted if it has been elapsed for =12 months prior to disease progression.
2. Prior treatment with EGFR targeting small molecules or antibodies.
3. Major surgery within 4 weeks of study treatment.
4. Brain metastases.
5. Meningeal carcinomatosis.
6. Known pre-existing interstitial lung disease (ILD).
7. Patients with a significant disease other than lung cancer; a significant disease is defined as a disease which, in the opinion of the investigator, may:

   * put the patient at risk because of participation in the study
   * influence the results of the study
   * cause concern regarding the patient's ability to participate in the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who has taken 30 mg Afatinib as initial dose and still on treatment for less than 28 days
Sampling Method: Non-Probability Sample
Enrollment: 69 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival rate | 6 months
  To assess the effect of afatinib 30 mg daily at the Investigator's discretion on progression-free survival rate (PFSR) at month 6.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationa University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tan DS, Yom SS, Tsao MS, Pass HI, Kelly K, Peled N, Yung RC, Wistuba II, Yatabe Y, Unger M, Mack PC, Wynes MW, Mitsudomi T, Weder W, Yankelevitz D, Herbst RS, Gandara DR, Carbone DP, Bunn PA Jr, Mok TS, Hirsch FR. The International Association for the Study of Lung Cancer Consensus Statement on Optimizing Management of EGFR Mutation-Positive Non-Small Cell Lung Cancer: Status in 2016. J Thorac Oncol. 2016 Jul;11(7):946-63. doi: 10.1016/j.jtho.2016.05.008. Epub 2016 May 23. PMID 27229180
- [Result] Sequist LV, Yang JC, Yamamoto N, O'Byrne K, Hirsh V, Mok T, Geater SL, Orlov S, Tsai CM, Boyer M, Su WC, Bennouna J, Kato T, Gorbunova V, Lee KH, Shah R, Massey D, Zazulina V, Shahidi M, Schuler M. Phase III study of afatinib or cisplatin plus pemetrexed in patients with metastatic lung adenocarcinoma with EGFR mutations. J Clin Oncol. 2013 Sep 20;31(27):3327-34. doi: 10.1200/JCO.2012.44.2806. Epub 2013 Jul 1. PMID 23816960
- [Result] Yang JC, Wu YL, Schuler M, Sebastian M, Popat S, Yamamoto N, Zhou C, Hu CP, O'Byrne K, Feng J, Lu S, Huang Y, Geater SL, Lee KY, Tsai CM, Gorbunova V, Hirsh V, Bennouna J, Orlov S, Mok T, Boyer M, Su WC, Lee KH, Kato T, Massey D, Shahidi M, Zazulina V, Sequist LV. Afatinib versus cisplatin-based chemotherapy for EGFR mutation-positive lung adenocarcinoma (LUX-Lung 3 and LUX-Lung 6): analysis of overall survival data from two randomised, phase 3 trials. Lancet Oncol. 2015 Feb;16(2):141-51. doi: 10.1016/S1470-2045(14)71173-8. Epub 2015 Jan 12. PMID 25589191